CLINICAL TRIAL: NCT02356601
Title: Lumbar Neuraxial Ultrasound Corrrelation With MRI
Status: Completed | Type: Observational
Sponsor: The Adelaide and Meath Hospital (Other)
Responsible Party: Principal Investigator, Karthikeyan Kallidaikurichi Srinivasan, Specialist Registrar,Anaesthetics, The Adelaide and Meath Hospital
Other Study IDs: 2013/03/20 chairman's action
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Ultrasound Imaging of Lumbar Spine
Keywords: MRI; Lumbar spine; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ultrasound is used increasingly to aid placement of neuraxial blocks. Good visibility of ligamentum duramater complex and posterior longitudinal ligament (LF, PLL) has a positive predictive value of 85% for successful neuraxial block. Dural puncture could still be feasible despite the absence of a good view, as reflected by a negative predictive value of 30%.

Poor neuraxial ultrasound view could be due to limitations of ultrasound or various other anatomical reasons which might include absent LF, calciﬁcation of ligaments, spinous process contact and presence or absence of epidural or subdural fat. This will be the first study of its kind to compare neuraxial ultrasound with MRI. The aim of this study is to look for anatomical correlation between neuraxial ultrasound and MRI at various lumbar interspinous levels and to look at factors that contribute to abnormal neuraxial imaging. Assuming the predicted abnormal ultrasound images to be around 30% and predicted abnormal MRI images to be 5%, 79 images should give a power of 0.9 and alpha 0.01 to analyse the association between the two. Sample Size Calculations were performed using statistical software R version 2.15.2

DETAILED DESCRIPTION:
After ethical committee approval, 20 consenting patients scheduled for MRI lumbar spine were included in the study. Patients with previous spinal surgeries or with gross spinal deformities were excluded. In all patients ultrasound scanning of the lumbar interspinous spaces was performed with curvilinear 2-5 MHz Sonosite probe. At each lumbar interspinous level (L1-2 to L5-S1) the best possible transverse and paramedian oblique sagittal view was obtained. The obtained ultrasound images were the graded based on the visibility of LF and PLL. The lumbar spine MRI images were analyzed by radiologists who were blinded to the ultrasound images. On MRI various parameters such as depth of epidural space, absence of LF, thickness of LF, characteristics of muscular and intervening fatty tissue, epidural/subdural fat thickness etc was noted. The correlation between neuraxial ultrasound images and various parameters observed in MRI was identified.

ELIGIBILITY:
Inclusion Criteria:

Any adult having MRI lumbar spine done

Exclusion Criteria:

Patients with previous spinal surgery Gross spinal deformities BMI more than 50

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having MRI lumbar spine done
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Association between abnormal MRI and poor view in Ultrasound | 2 hour post completion of MRI
  Ultrasound images were the graded based on the visibility of Ligamentum Flavum (LF) and Posterior longitudinal ligament (PLL) as good (Both PLL and LF visible), intermediate (either LF or PLL only visible) or poor (both LF and PLL not visible. An abnormal MRI is defiined as one with any of the following - presence of fascet joint hypertrophy or non fusion of ligamentum flavum.